CLINICAL TRIAL: NCT06332014
Title: A Phase 4 Single Arm Open Label Study for the Efficacy and Safety of Prolia in Treatment of Male Subjects With Osteoporosis in Mainland China
Brief Title: Evaluation of Efficacy and Safety of Prolia in Subjects of Male Osteoporosis in Mainland China
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20210123
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Osteoporosis
Keywords: Prolia; Denosumab; AMG 162; Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Denosumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolia (Experimental): Participants will receive Prolia every six months (Q6M)
  Interventions: Drug: Prolia

INTERVENTIONS:
Drug: Prolia — Partcipants will receive subcutaneous (SC) injections of Prolia Q6M.
  Other Names: Denosumab

SUMMARY:
The primary objective of this study is to evaluate the efficacy of Prolia on lumbar spine BMD at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory Chinese men aged ≥ 30 years and ≤ 90 years old at the time of signing the informed consent.
* Men at the time of screening will be required to have lumbar spine or total hip BMD T-score ≤ -2.5 or T-score ≤ -1.5 and a history of a fragility fracture.
* Have to have at least two intact vertebrae at baseline (L1-L4).

Exclusion Criteria:

* Any condition that could affect bone metabolism such as Paget's disease of bone, osteomalacia including secondary causes of osteoporosis (subjects with low testosterone levels are allowed).
* Hyper- or hypothyroidism; however, stable subjects, in the investigator's opinion, on thyroid hormone replacement therapy are allowed.
* Participants with a history of any cancer (cured basal cell or squamous cell cancers are allowed).
* Any condition that in the opinion of the investigator would not allow the subject to complete 1 year study and comply with the requirement of the study protocol.
* Hypogonadism requiring testosterone replacement therapy unless on a stable dose for at least 12 months.
* Administration of intravenous bisphosphonate, or fluoride (except for dental treatment) or strontium ranelate. Systemic glucocorticoids: ≥ 7.5 mg prednisone equivalent per day for more than 14 days within 3 months before randomization. Any bone anabolic treatment within 1 year. Anabolic steroids or testosterone: any use within 6 months before randomization.
* Oral bisphosphonates treatment.
* Known to have tested positive for human immunodeficiency virus, hepatitis C virus, hepatitis B surface antigen, or cirrhosis of the liver.
* Received any solid organ or bone marrow transplant or is on chronic immunosuppression for any reason.
* Oral/dental conditions that would require an intervention including tooth extraction during the course of the study and invasive dental work (per local oral surgeon's assessment) planned in the next 12 months.
* Any prior use of products containing denosumab.
* Currently receiving treatment in another investigational device or drug study, or less than 1 month since ending treatment on another investigational device or drug study(ies). Other investigational procedures while participating in this study are excluded.
* Vitamin D levels < 20 ng/mL (subjects are allowed into the study after vitamin D levels are corrected and subjects re-screened).
* Albumin-adjusted serum calcium levels < 8.5 mg/dl or > 10.5 mg/dl.

Ages: 30 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 102 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2027-01-23 (Estimated); Study Completion 2027-01-23 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in bone mineral density (BMD) of lumbar spine at month 12 | Baseline and Month 12

SECONDARY OUTCOMES:
Percent change from baseline in serum C-terminal telopeptide (CTx) at month 3, 6, 9, and 12 | Baseline and Months 3, 6, 9, and 12
Percent change from baseline in serum procollagen Type 1 N-Telopeptide (P1NP) at month 3, 6, 9, and 12 | Baseline and Months 3, 6, 9, and 12
Percent change from baseline in total hip and femoral neck BMD at month 6 and 12 | Baseline and Months 6 and 12
Percent change from baseline in lumbar spine BMD at month 6 | Baseline and Month 6
Number of participants with adverse events (AE) | Up to 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (16):
- China (16):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Jishuitan Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Sun Yat-sen Memorial Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - The Fourth Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Huaian First Peoples Hospital, Huaian, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Peoples Hospital of Kunshan, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Jiangxi Provincial Peoples Hospital, Nanchang, Jiangxi
  - Pingxiang Peoples Hospital, Pingxiang, Jiangxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanghai Sixth Peoples Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com